CLINICAL TRIAL: NCT04559932
Title: Paediatric Chronic Tracheostomy Care: An Evaluation of an Innovative Competency-based Education Program for Community Health Care Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Reshma Amin, Associate Professor, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1000057879
Record Dates: First submitted 2020-08-27; First posted 2020-09-23 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Evaluation of HomeCare RN Respiratory Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The knowledge and self-efficacy pre-tests will be completed at the start of the course and the post-test will be completed after the course at the end of the day. Study participants will complete tests independently using paper and pencil. Six weeks and six months post course completion, the knowledge and self-efficacy tests will be completed using REDcap (Research Electronic Data Capture), a secure web application for building and managing online surveys and databases or via telephone as per participant preference. Study participants will be sent a link to complete the tests online for the subsequent study visits. Study participants will receive 2 reminder emails (1 week apart) and 1 reminder phone call after the email reminders (if applicable) to complete the tests. Monthly telephone calls by the RA will be made to review the HCP experience logs.
  Interventions: Other: Tracheostomy Training Course
- Control (No Intervention): Study participants in the control arm will be offered complementary attendance in the Health Tech Junior enterostomy and vascular access competency based training course while awaiting their session. This is being done to minimize the potential confound of generalized improvements in self-efficacy that may occur as a result of participating in an 8 hour learning opportunity at SickKids. The control group will also complete the tracheostomy course during session 3 and 4 but this will occur outside the window of data collection for the study procedures. Data collection intervals as described above for the intervention group will be followed for the control group.

INTERVENTIONS:
Other: Tracheostomy Training Course — A standardized competency-based education tracheostomy module has been developed by the investigator group in collaboration with Respiratory Medicine, Complex Care, Respiratory Therapy, Nursing Education, Family Advisory Network and the Learning Institute at SickKids. Instructional methods for the full module are based on principles of adult learning and evidence from the procedure education literature and include the use of interactive, small-group teaching, hands-on simulation-based learning stations with relevant equipment as well as a formal assessment of knowledge and skills using simulation. Pre-learning packages are sent to course attendees at the time of registration to facilitate higher level discussions on the day of the course. While investigators have rigorously developed the curriculum and evaluation measures, the course outcomes remain unknown.
  Arms: Intervention

SUMMARY:
This project will evaluate a new course developed for nurses that provide care to children with breathing technology including breathing tubes and home breathing machines. The investigators plan to assess the nurses' knowledge and comfort of their ability to care for these medical technologies prior to the course as well as their ability to retain their knowledge 6 weeks and 6 months after course completion.

DETAILED DESCRIPTION:
A structured program evaluation considering a hierarchy of outcomes is essential to determine whether the tracheostomy module is associated with improved knowledge and skills for CHPs (community health providers). This investigators proposed study is guided by the evaluation of knowledge acquisition and self-efficacy as a theoretical framework 24. CHPs' sense of self-efficacy or perceived capability in caring for this population is important to foster to potentially mitigate significant morbidity and mortality, while ultimately striving for safe, high-quality clinical care for these medically complex children.

ELIGIBILITY:
Inclusion Criteria:

* Course registrants for the competency-based tracheostomy education course from VHA Home Healthcare agency
* Consent to study participation
* English speaking

Exclusion Criteria:

• Previously attended the competency-based tracheostomy course at SickKids

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The difference in the immediate knowledge retention scores of tracheostomy course participants versus controls at 6 week follow-up | 6 weeks
  Knowledge Assessment - Tracheostomy Tubes: Multiple choice question (MCQ) tests have been developed by clinical experts. These tests focus on the important knowledge required to care for a child with a tracheostomy tube. Major themes include: i) clinical assessment; ii) safety; iii) general care; iv) troubleshooting/ emergency management. Higher Scores mean better knowledge retention.

SECONDARY OUTCOMES:
The difference in the sustained knowledge retention scores of course participants versus controls at 6 month follow-up | 6 weeks and 6 months
  Knowledge Assessment - Tracheostomy Tubes: Multiple choice question (MCQ) tests have been developed by clinical experts. These tests focus on the important knowledge required to care for a child with a tracheostomy tube. Major themes include: i) clinical assessment; ii) safety; iii) general care; iv) troubleshooting/ emergency management. Higher Scores mean better knowledge retention.
The difference in the self-efficacy scores of course participants versus controls at 6 weeks and 6 month follow-up | 6 weeks and 6 months
  Self-Efficacy - Tracheostomy Tubes: A self-efficacy survey that is content relevant for tracheostomy tubes has been developed based on Bandura's framework 24. The survey consists of 16 items assessing the registrants' perceived capability to perform each aspect of care on a likert scale with a 0-100 response interval. Higher Scores mean more self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi JY, Orkin J, Walsh CM, Chu S, Keilty K, McKay S, Mocanu C, Qazi A, Ambreen M, Amin R. Pediatric Chronic Tracheostomy Care: An Evaluation of an Innovative Competency-Based Education Program for Community Health Care Providers. Front Pediatr. 2022 May 31;10:885405. doi: 10.3389/fped.2022.885405. eCollection 2022. PMID 35757113